CLINICAL TRIAL: NCT02229344
Title: Cohort Study of Newly Diagnosed Moderate to Severe Ulcerative Colitis in Tertiary Referral Hospital Setting in Korea
Brief Title: Study of Clinical Course of Newly Diagnosed Moderate to Severe Ulcerative Colitis in Korea
Acronym: MOSAIK
Status: Completed | Type: Observational
Sponsor: Janssen Korea, Ltd., Korea (Industry)
Responsible Party: Sponsor
Other Study IDs: CR103116; REMICADECRD4016 (Other: Janssen Korea, Ltd., Korea); INF-KOR-5005 (Other: Janssen Korea, Ltd., Korea)
Record Dates: First submitted 2014-08-28; First posted 2014-09-01 (Estimated); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Colitis, Ulcerative
Keywords: colitis, ulcerative; MOSAIK; REMICADE; Infliximab
MeSH Terms: conditions — Colitis, Ulcerative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood sample will be collected and stored for genetic and biomarker research from participants who agree to give additional informed consent form.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Newly Diagnosed Moderate to Severe Ulcerative Colitis: Participants with newly diagnosed moderate to severe ulcerative colitis in a tertiary referral hospital within 4 weeks before prior to enrollment will be observed.
  Interventions: Other: No Intervention

INTERVENTIONS:
Other: No Intervention — Participants with newly diagnosed moderate to severe ulcerative colitis in a tertiary referral hospital within 4 weeks before prior to enrollment will be observed.

SUMMARY:
The purpose of this study is to describe clinical course of newly diagnosed moderate to severe ulcerative colitis (chronic inflammatory disease of the colon) in tertiary referral hospitals in Korea for 5-year follow-up under usual care.

DETAILED DESCRIPTION:
This is a multicenter (when medical research study takes place in more than one country), prospective (study following participants forward in time), disease-oriented and hospital-based 5-year follow-up longitudinal study in Korean participants with newly diagnosed moderate to severe ulcerative colitis who visit tertiary referral hospital. As the study is observational in nature, no intervention will be received by participants. Efficacy will primarily be assessed by number of relapses and percentage of participants achieving sustained remission (clinical, endoscopic and combined remission).

ELIGIBILITY:
Inclusion Criteria:

* Participant is newly diagnosed with moderate to severe ulcerative colitis in a tertiary referral hospital within 4 weeks prior to enrollment
* The diagnosis was based on symptoms consistent with ulcerative colitis lasting for more than 4 weeks, excluding infections and other acute or chronic non-infectious bowel syndrome conditions
* Participants meet diagnostic criteria for ulcerative colitisif at least 3 out of 4 of the following are met: 1) A History of diarrhea and/or blood/pus in stool, 2) Macroscopic appearance at endoscopy, with continuous mucosal inflammation affecting the rectum in continuity with some or all of the colon, 3) Microscopic features on biopsy consistent with ulcerative colitis, 4) No suspicion of Crohn's disease or indeterminate colitis
* Participants are willing to participate in regular follow-up visits
* Participant is willing to participate in the study and has signed the informed consent

Exclusion Criteria:

* Participants in an interventional clinical trial with systemic corticosteroid, biologics (including, but not limited to, infliximab, golimumab, adalimumab and vedolizumab, etc) and other drugs (sulfasalazine, medalamine, azathioprine, tofacitinib, etc) for ulcerative colitis
* Having experienced colectomy such as subtotal colectomy with ileorectostomy or colectomy with ileoanal pouch, Koch pouch, or ileostomy for ulcerative colitis, or planning surgical treatment within 1 year from enrollment
* A current diagnosis of indeterminate colitis, or current diagnosis or history of Crohn's disease

Min Age: 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Participants with newly diagnosed moderate to severe ulcerative colitis in a tertiary referral hospital within 4 weeks before prior to enrollment will be observed.
Sampling Method: Non-Probability Sample
Enrollment: 368 (Actual)
Dates: Start 2014-07-01 (Actual); Primary Completion 2022-02-22 (Actual); Study Completion 2022-02-22 (Actual)

PRIMARY OUTCOMES:
Total Number of Relapses in Year 1 | Year 1
  Relapse is defined as increase in Mayo or partial Mayo score of more than or equal to (>=) 3 points from clinical response or remission. Mayo score is a discrete ordinal scale with total score ranging from 0 (normal or inactive disease) to 12 (severe disease) and partial Mayo score ranges from 0 (normal or inactive disease) to 9 (severe disease). Relapses will be categorized as: infrequent (less than or equal to [<=] 1 relapse per year), frequent pattern (>=2 relapses per year) and continuous (persistent symptoms of active ulcerative colitis without a period of remission).
Total Number of Relapses in Year 3 | Year 3
  Relapse is defined as increase in Mayo or partial Mayo score of >=3 points from clinical response or remission. Mayo score is a discrete ordinal scale with total score ranging from 0 (normal or inactive disease) to 12 (severe disease) and partial Mayo score ranges from 0 (normal or inactive disease) to 9 (severe disease). Relapses will be categorized as: infrequent (<=1 relapse per year), frequent pattern (>=2 relapses per year) and continuous (persistent symptoms of active ulcerative colitis without a period of remission).
Total Number of Relapses in Year 5 | Year 5
  Relapse is defined as increase in Mayo or partial Mayo score of >=3 points from clinical response or remission. Mayo score is a discrete ordinal scale with total score ranging from 0 (normal or inactive disease) to 12 (severe disease) and partial Mayo score ranges from 0 (normal or inactive disease) to 9 (severe disease). Relapses will be categorized as: infrequent (<=1 relapse per year), frequent pattern (>=2 relapses per year) and continuous (persistent symptoms of active ulcerative colitis without a period of remission).
Percentage of Participants With Sustained Remission in Year 1 | Year 1
  Clinical remission is <=2 points with no individual sub-score >1 point using total or partial Mayo Score. Mayo score is a discrete ordinal scale with total score ranging from 0 (normal or inactive disease) to 12 (severe disease) and partial Mayo Score score ranges from 0 (normal or inactive disease) to 9 (severe disease).
Percentage of Participants With Sustained Remission in Year 3 | Year 3
  Clinical remission is <=2 points with no individual sub-score >1 point using total or partial Mayo Score. Mayo score is a discrete ordinal scale with total score ranging from 0 (normal or inactive disease) to 12 (severe disease) and partial Mayo Score score ranges from 0 (normal or inactive disease) to 9 (severe disease).
Percentage of Participants With Sustained Remission in Year 5 | Year 5
  Clinical remission is <=2 points with no individual sub-score >1 point using total or partial Mayo Score. Mayo score is a discrete ordinal scale with total score ranging from 0 (normal or inactive disease) to 12 (severe disease) and partial Mayo Score score ranges from 0 (normal or inactive disease) to 9 (severe disease).

SECONDARY OUTCOMES:
Mean Time to Relapse | Year 1, 3 and 5
  Relapse is defined as increase in mayo or partial Mayo score of more than or equal to (>=) 3 points from clinical response or remission. Mayo score is a discrete ordinal scale with total score ranging from 0 (normal or inactive disease) to 12 (severe disease) and partial Mayo score ranges from 0 (normal or inactive disease) to 9 (severe disease). Average time taken to occurrence of first relapse will be observed.
Percentage of Participants With Sustained Clinical Response | Year 1, 3 and 5
  Response is defined as decrease in Mayo or partial Mayo score of >=3 points from Baseline and decrease in Mayo score of >=30 percent (%) from Baseline and decrease in the rectal bleeding score >=1 or an absolute rectal bleeding score of 0 or 1.
Total Number of Ulcerative Colitis-Related Hospitalizations | Year 3 and 5
  Total number of ulcerative colitis-related hospitalizations will be observed.
Total Days of Ulcerative Colitis-Related Hospitalizations | Year 3 and 5
  Total days of ulcerative colitis-related hospitalizations will be observed.
Percentage of Participants With Colectomy | Year 3 and 5
  Percentage of participants who will be going for surgery to remove part or all of the colon will be observed.
Percentage of Participants With Death | Year 3 and 5
  Percentage of participants with death (ulcerative colitis related and non-ulcerative colitis related) will be observed.
Mean Change From Baseline in Disease Extent at Year 1, 3 and 5 | Baseline, Year 1, 3 and 5
  Colonoscopy (a medical examination of the colon by a physician using a colonoscope) will be conducted to explore the extent of lesion to determine extent of disease.
Mean Change From Baseline in Inflammatory Bowel Disease Questionnaire (IBDQ) Score at Year 1, 3 and 5 | Baseline and Year 1, 3 and 5
  The IBDQ evaluates the effect of the participants' inflammatory bowel disease on the quality of life Scores range from 32 to 224 with higher scores indicating better quality of life.
Mean Change From Baseline in Short Form Survey (SF 12) Score at Year 1, 3 and 5 | Baseline, Year 1, 3 and 5
  The SF12 is a generic measure physical and mental health, it is is weighted and summed to provide easily interpretable scales. Physical and Mental Health Composite Scores (PCS & MCS) are computed using the scores of twelve questions and range from 0 to 100, where a zero score indicates the lowest level of health measured by the scales and 100 indicates the highest level of health.
Change From Baseline in Hospital Anxiety and Depression Scale (HADS) Score at Year 1, 3 and 5 | Baseline, Year 1, 3 and 5
  The HADS is a self-assessment scale for the symptom severity of anxiety disorders and depression. It comprises of 14 items, and each item is rated on a four-point scale (0-3). All seven answers are summarized and calculated to a total score to the anxiety scale and to the depression scale with a maximum score of 21 points for each scale.
Percentage of Participants Treated With Immune Modulators, Systemic Steroids and Biologics | Baseline up to Year 5
  Percentage of participants treated with immune modulators (azathioprine or 6-mercaptoprine at least a consecutive 3-month course), systemic steroids and biologics will be reported.
Mean Time to First Treatment With Immune Modulators, Systemic Steroids and Biologics From Baseline | Baseline up to Year 5
  Time to first administration of immune modulators like azathioprine or 6-mercaptoprine for at least a consecutive 3-month course, systemic steroids and biologics from Baseline will be observed.
Number of Participants With Complementary and Alternative Medicine (CAM) use and Satisfaction | Baeline up to Year 5
  Number of participants with CAM use and satisfaction will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Korea, Ltd., Korea Clinical Trial, Study Director — Janssen Korea, Ltd., Korea
Locations (15):
- South Korea (15):
  - Ansan-si
  - Busan
  - Cheonan
  - Cheongju-si
  - Daegu
  - Daejeon
  - Guri-si
  - Gwangju
  - Iksan
  - Incheon
  - Kwanju
  - Seongnam-si
  - Seoul
  - Suwon
  - Wŏnju